CLINICAL TRIAL: NCT03136354
Title: Prospective Randomized Trial Comparing Endoscopic Submucosal Dissection Against Laparoscopic Assisted Gastrectomy for Treatment of Early Gastric Cancer
Acronym: LGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Philip Wai Yan Chiu, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2009.165T
Record Dates: First submitted 2016-11-27; First posted 2017-05-02 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Early Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ESD Group (Active Comparator): Endoscopic Submucosal Dissection
  Interventions: Procedure: Endoscopic Submucosal Dissection
- LAG Group (Active Comparator): Laparoscopic Assisted Gastrectomy
  Interventions: Procedure: Laparoscopic assisted Gastrectomy

INTERVENTIONS:
Procedure: Endoscopic Submucosal Dissection
  Arms: ESD Group
Procedure: Laparoscopic assisted Gastrectomy
  Arms: LAG Group

SUMMARY:
The investigators compared the perioperative, oncological, functional and immunological outcomes of endoscopic submucosal dissection against laparoscopic assisted gastrectomy for treatment of early gastric cancer. With virtually no abdominal incisions and minimal pain induced, endoscopic submucosal dissection is expected to be less invasive when compared to laparoscopic assisted gastrectomy for treatment of early gastric cancer. This study will show that endoscopic submucosal dissection is associated with a significantly better perioperative recovery and less immunological disturbance. Moreover, it will also induce a better long term outcomes as the stomach can be preserved, hence the digestive function is maintained to prevent long term functional morbidities of the gastrointestinal tract.

This study will be the unique first study in the literature to show that intramucosal early gastric cancer can be adequately treated by endoscopic submucosal dissection with better perioperative, functional and quality of life outcomes when compared to laparoscopic assisted gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Early gastric cancer with biopsy confirmed high grade dysplasia or adenocarcinoma (intestinal type)
2. Preoperative investigation with magnifying endoscopy and / or EUS predicted to be mucosal lesion
3. Any tumor size if the early gastric cancer has no ulceration
4. Tumor size ≤ 3cm if the early gastric cancer has ulceration

Exclusion Criteria:

1. Gastric cancer with preoperative magnifying endoscopy and / or EUS predicted to beyond submucosal invasion
2. Poorly differentiated or signet ring cell adenocarcinoma
3. Age > 80 or < 16
4. Pregnancy
5. ASA > IV

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-05; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Complication | 30 days after procedure

SECONDARY OUTCOMES:
Postop VAS score on pain measurement | 30 days
  Measured by VAS pain score daily until the day of discharge by dedicated independent assessor Daily measurement until the day of discharge the type and dose of analgesic requirement is also documented
Hospital stay | through study completion, an average of 1 year
  The number of days that patient stayed in hospital
Time (hours) for Operative | Up to 24 hours
  The Time measured by hours from start of operation after general anesthesia until end of the operation
Quality of life assessment by SF36 | From date of operation on every followup appointment until 24 months after operation
  As measured by SF 36
Mortality | 30 days after procedure
Overall Survival | up to 5 years after operation
Recurrence | up to 5 years after operation
Disease free survival | up to 5 years after operation

CONTACTS AND LOCATIONS:
Overall Officials: Philip W Chiu, MD, FRCSEd, Principal Investigator — Dept of Surgery, The Chinese University of Hong Kong
Locations (1):
- Combined Endoscopy Center, Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No